CLINICAL TRIAL: NCT04411160
Title: Comparative Study Between the Effect of Vitamin C vs. Nitric Oxide in Weaning of Patients With Prolonged Ventilation Due to ARDS
Brief Title: Vitamin C Versus Nitric Oxide in Prolonged Ventilation
Status: Completed | Type: Observational
Sponsor: King Abdul Aziz Specialist Hospital (Network)
Responsible Party: Sponsor
Other Study IDs: ICU-32-20
Record Dates: First submitted 2020-05-21; First posted 2020-06-02 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: ARDS
MeSH Terms: interventions — Ascorbic Acid; Nitric Oxide; Ventilators, Mechanical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Group A: Patients of group A received inhalation of nitric oxide stared by 50 parts/billion(ppb) as starting dose titrated according to patient's saturation reaching to 90 ppb as a maximum dose.
  Interventions: Drug: Nitric Oxide; Device: ventilators
- Group B: While patients of group B received 4 gram of vitamin c slowly intravenous once daily for 4 days duration.
  Interventions: Drug: Vitamin C; Device: ventilators

INTERVENTIONS:
Drug: Vitamin C — 4 gram of vitamin c slowly intravenous once daily for 4 days duration.
  Groups: Group B
Drug: Nitric Oxide — nitric oxide stared by 50 parts/billion(ppb) as starting dose titrated according to patient's saturation reaching to 90 ppb as a maximum dose
  Groups: Group A
Device: ventilators — All selected patients received conventional ventilation with protective lung strategy for 10 days with Controlled mechanical ventilation mode(CMV), fraction inspired oxygen (FIO2) of 100%, Positive end expiratory pressure(PEEP) of 10 cm H2O or more to achieve target arterial oxygen saturation(SPO2) of 90%

SUMMARY:
This a prospective double-blind study done in King Abdul-Aziz specialist hospital between January 2019 and April 2020 in the intensive care unit on 60 patients with difficult weaning and ventilated for 10 days. Allocated randomly in two groups 30 patients in each. All patients in both groups continued on the same conventional ventilation but Group A received nitric oxide (NO) while group B received vitamin C intravenous. The duration of the study last 16 days. during this period, APCHII score, Hemodynamics, Chest Xray, hypoxic index, lung compliance, Recruitment maneuver, arterial blood saturation, LDH, C-reactive protein used as indicator for improvement. Number of patients weaned from the ventilator and patients died also recorded.

DETAILED DESCRIPTION:
All selected patients received conventional ventilation with protective lung strategy for 10 days with Controlled mechanical ventilation mode(CMV), fraction inspired oxygen (FIO2) of 100%, Positive end expiratory pressure(PEEP) of 10 cm H2O or more to achieve target arterial oxygen saturation(SPO2) of 90% or more with sedation by midazolam infusion to achieve Richmond Agitation- Sedation Scale (RASS) -2 to -3 and fentanyl infusion for pain control between 50-100 mg/min. Protective lung strategy was strictly applied in form of head elevation more than 30°, broad spectrum antibiotics according to our antibiotic regimen, daily assessment for both analgesic and sedative dose were given to patients, early naso-gastric feeding started to prevent ventilator associated pneumonia and daily trial was done to reduce PEEP to prevent more lung injury from ventilation also qualitative sputum culture was taken after one week from ventilation. After 10 days from the conventional ventilation those who could not be weaned from the ventilator and still had the former criteria mentioned before (Uncompensated hypercapnia with PH<7.25, and/or Hypoxic index less than 200) included in our study. Percutaneous dilatation tracheostomy done for all patients in both groups. 60 patients randomly allocated in 2 groups. Randomization sequence was created using Excel 2007 (Microsoft, Redmond, WA, USA) with a 1:1 allocation using random block sizes of 2 and 4 by an independent doctor. In this way, sequence generation and type of randomization can be expressed at the same time. Each group included 30 patients. Patients of group A received inhalation of nitric oxide stared by 50 parts/billion(ppb) as starting dose titrated according to patient's saturation reaching to 90 ppb as a maximum dose. While patients of group B received 4 gram of vitamin c slowly intravenous once daily for 4 days duration. Improvement of general condition of the patients monitored in our study by APACH II score and core body temperature. improvement of the lungs condition monitored in our study clinically by monitoring: oxygen saturation, hypoxic index, compliance and response to recruitment maneuver ( Recruitment maneuver is considered clinical test of lung compliance and start by increase the peak inspiratory pressure to 40 cm/H2O for 40 sec and observe the saturation (SpO2) if improved to more than 95% considered responder in our study).(18) and radiologically by size of parenchymatous lung infiltration on chest X ray. The duration of the study 16 days

ELIGIBILITY:
Inclusion Criteria:

* ARDS

Exclusion Criteria:

* systemic disease as diabetes and hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — adult only
Study Population: This a prospective cohort study done in King Abd el Aziz specialist hospital between January 2019 and April 2020 in the intensive care unit on 60 patients with respiratory failure and showed failure of weaning from ventilator either due to medical or surgical causes. King Abdelaziz research and ethical committee approved the project.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-04-19 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
tissue oxygenation | 2 weeks
  observe the arterial oxygen saturation SpO2

CONTACTS AND LOCATIONS:
Locations (1):
- King abd el Aziz specialist hospital, Ta'if, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No